CLINICAL TRIAL: NCT07057362
Title: Effect of Vitamin D Deficiency on the Frequency and Severity of Spinal Anesthesia-Induced Hypotension in Pregnant Women Undergoing Cesarean Section
Status: Recruiting | Type: Observational
Sponsor: Duzce University (Other)
Responsible Party: Sponsor
Other Study IDs: 2025/63
Record Dates: First submitted 2025-06-30; First posted 2025-07-09 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Spinal Anesthesia-induced Hypotension; Vitamin D Deficiency; Cesarean Section
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Vitamin D Deficient Group: Pregnant women with serum 25-hydroxyvitamin D levels below the defined deficiency threshold
  Interventions: Other: Intraoperative Hemodynamic Monitoring
- Vitamin D Sufficient Grup: Pregnant women with normal or sufficient vitamin D levels
  Interventions: Other: Intraoperative Hemodynamic Monitoring

INTERVENTIONS:
Other: Intraoperative Hemodynamic Monitoring — Continuous intraoperative monitoring of systolic blood pressure and heart rate following spinal anesthesia. Vasopressor usage and total fluid administration will be recorded.

SUMMARY:
Spinal anesthesia-induced hypotension remains a common and significant complication during cesarean sections, posing risks for both mother and fetus. Vitamin D deficiency, frequently observed in pregnant women, is associated with altered vascular function and potential hemodynamic instability. This prospective observational study aims to investigate whether vitamin D deficiency is associated with an increased incidence and severity of spinal anesthesia-induced hypotension in pregnant women undergoing elective cesarean delivery. Vitamin D levels will be measured preoperatively, and intraoperative hemodynamic parameters will be closely monitored. The findings could contribute to improved management strategies for pregnant patients at risk of severe hypotension.

DETAILED DESCRIPTION:
Detailed Description Spinal anesthesia is the most commonly used technique for cesarean section and is associated with a high incidence of maternal hypotension, which can adversely affect both maternal well-being and neonatal outcomes. Despite standard preventive strategies such as fluid preloading and vasopressor use, significant hypotension still occurs in a considerable proportion of patients.

Vitamin D deficiency is a prevalent condition among pregnant women and has been implicated in the modulation of cardiovascular and autonomic functions. Low serum levels of 25-hydroxyvitamin D may impair vascular smooth muscle contractility, endothelial function, and baroreflex sensitivity, potentially contributing to exaggerated hypotensive responses under spinal anesthesia.

This prospective observational study aims to evaluate the relationship between maternal vitamin D status and the incidence and severity of spinal anesthesia-induced hypotension during elective cesarean delivery. Eligible pregnant women scheduled for elective cesarean section under spinal anesthesia will have their serum 25-hydroxyvitamin D levels measured preoperatively. Intraoperative hemodynamic parameters will be continuously monitored, and episodes of hypotension will be recorded and analyzed in relation to vitamin D status.

The primary outcome of the study is the incidence of spinal hypotension, defined as a ≥20% decrease in systolic blood pressure from baseline or an absolute value below 90 mmHg. Secondary outcomes include total vasopressor dose, fluid requirement.

Findings from this study may identify vitamin D deficiency as a novel risk factor for spinal anesthesia-induced hypotension and inform new preventive strategies for hemodynamic management in cesarean deliveries

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged 18 years or older
* Scheduled for elective cesarean delivery under spinal anesthesia
* Able and willing to provide written informed consent

Exclusion Criteria:

* Emergency cesarean sections
* History of significant cardiovascular disease (e.g., arrhythmia, heart failure)
* Known neurological disorders affecting autonomic function
* Current vitamin D supplementation within the past 30 days
* Inability to undergo blood sampling or provide valid hemodynamic data
* Contraindication to spinal anesthesia

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Pregnant women aged 18 years and older who are scheduled for elective cesarean section under spinal anesthesia at a tertiary care university hospital. All participants will be clinically stable and provide informed consent prior to enrollment. The study population will be stratified based on serum vitamin D levels into deficient and sufficient groups for analysis of hypotension outcomes.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-12-30 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Hypotension After Spinal Anesthesia | ntraoperative (0-30 minutes after spinal anesthesia)
  Hypotension is defined as a ≥20% decrease in systolic blood pressure from baseline or an absolute systolic value <90 mmHg. The presence or absence of hypotension will be recorded.

SECONDARY OUTCOMES:
Total Vasopressor Dose Administered | Intraoperative (0-30 minutes after spinal anesthesia)
  Cumulative amount (in mg) of vasopressor (e.g., ephedrine or phenylephrine) used to manage hypotension.
Total Crystalloid Volume Administered | Intraoperative (0-30 minutes after spinal anesthesia)
  Total amount (in mL) of intravenous crystalloids given from the time of spinal anesthesia until delivery.

CONTACTS AND LOCATIONS:
Locations (1):
- Duzce University Faculty of Medicine, Department of Anesthesiology and Reanimation, Düzce, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The study involves sensitive clinical data from pregnant women. Individual participant data will not be shared publicly due to privacy concerns.